CLINICAL TRIAL: NCT03511313
Title: A Prospective, Multi-centers, Randomized, Controlled Study of Assessing the Safety and Efficacy of Sterile Irrigated Deflectable Ablation Catheter Used in Renal Artery in Primary Hypertension
Brief Title: Renal Denervation With Sterile Irrigated Deflectable Ablation Catheter Used in Renal Artery in Primary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Synaptic Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNP-CT-1601
Record Dates: First submitted 2018-03-26; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Primary Hypertension
Keywords: Primary Hypertension; Renal Denervation
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renal denervation (Experimental): Renal angiography and renal denervation (with sterile irrigated deflectable ablation catheter in renal artery), and maintaining anti-hypertensive medications
  Interventions: Device: Renal denervation; Diagnostic Test: Renal angiography
- Renal angiography (Sham Comparator): Renal angiography and maintaining anti-hypertensive medications
  Interventions: Diagnostic Test: Renal angiography

INTERVENTIONS:
Device: Renal denervation — After a renal angiography according to standard procedures, subjects are treated with renal denervation (with sterile irrigated deflectable ablation catheter in renal artery), if without renal anatomic abnormality not detected by Renal CT/CTA.
  Other Names: Renal angiography
  Arms: Renal denervation
Diagnostic Test: Renal angiography — A renal angiography according to standard procedure.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of renal denervation with sterile irrigated deflectable ablation catheter used in renal artery in primary hypertension in China.

ELIGIBILITY:
Inclusion Criteria:

* Individual is ≥18 years and ≤65 years old.
* Primary hypertension.
* Screen criteria: Individual who received a stable anti-hypertensive medication regimen including 2 or more anti-hypertensive medications of different classes prior to screening, and at the initial screening visit, he has an office systolic blood pressure(SBP)≥ 150mmHg, and ≤180mmHg, is entering the screening period after writing the informed consent. Individual is receiving a 4week standard dose of amlodipine besylate (Norvasc) and Losartan Potassium and Hydrochlorothiazide tablets (HYZAAR®), and has a SBP≥150mmHg and<180mmHg at the second week after screening, and has an Ambulatory 24-hour daytime average systolic blood pressure monitoring ≥140mmHg and <170mmHg at the fourth week after screening.

Exclusion Criteria:

* Secondary hypertension.
* History of prior renal artery intervention including balloon angioplasty or stenting.
* Renal artery stenosis (≥50%) in either renal artery.
* Main renal arteries with <4mm, or >8mm in diameter.
* Main renal arteries with <20mm in length.
* Estimated glomerular filtration rate (eGFR) of <40 ml/(min•1.73m2).
* History of Stroke or TIA within 6 months prior to screening period.
* History of Acute coronary syndrome within 6 months prior to screening period.
* Structural heart disease without receiving effective treatment; Coronary heart disease with β blockers; severe peripheral artery disease that affecting blood pressure measurement and other unqualified conditions evaluated by investigator.
* Heart failure (NYHA classification Ⅲ-Ⅳ).
* Coagulation disorders associated with significant bleeding tendency, and history of other blood system diseases.
* History of cancer.
* Type 1 diabetes mellitus; Type 2 diabetes mellitus with target organ injuring.
* Acute or severe systemic inflammatory response syndrome.
* Any other serious medical condition unqualified to participate in this study evaluated by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in daytime average systolic blood pressure as measured by 24-hour Ambulatory Blood Pressure Monitoring | from baseline to 3 months post-procedure
  Primary effective outcome measure

SECONDARY OUTCOMES:
Change in office systolic blood pressure | from baseline to 3 months post-procedure
  Secondary effective outcome measure
Classes of anti-hypertensive medicine taken by participants | 6 months post-procedure
  Secondary effective outcome measure
Incidence of achieving target office systolic blood pressure (office SBP<140mmHg) | from 3 months post-procedure to 6 months post-procedure
  Secondary effective outcome measure

OTHER OUTCOMES:
Change in serum creatinine | from baseline to 3 months post-procedure and 6 months post-procedure
  Safety outcome assessment
Incidence of renal stenosis | 6 months post-procedure
  Safety outcome assessment
Other acute and chronic safety evaluating by the incidence of major adverse event | 6 months post-procedure
  Safety outcome assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yong Huo, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China